CLINICAL TRIAL: NCT00120783
Title: Efficacy and Tolerability of an Antiretroviral bi-Therapy in HIV-1 Infected Patients With Multidrug Resistant HIV ANRS 109 Vista Trial.
Brief Title: Efficacy and Tolerability of an Antiretroviral Bi-Therapy in HIV Infected Patients With Multidrug Resistance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 109 VISTA
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2007-01

CONDITIONS: HIV Infections
Keywords: Treatment Failure; HIV infections
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Ritonavir

INTERVENTIONS:
Drug: Indinavir
Drug: Lamivudine
Drug: Ritonavir

SUMMARY:
This study investigated whether a calibrated reduction in antiretroviral drug pressures could stabilize the evolution and the pathogenic potential of resistant HIV viruses.

DETAILED DESCRIPTION:
In patients with HIV multidrug resistance, maintaining a failing full-dose HAART regimen usually results in significant drug toxicity and in continued accumulation of resistance mutations that can preclude future therapeutic options. In contrast, treatment interruption provokes the reemergence of wild-type virus with full replicative and pathogenic capacity. The researchers investigated whether a calibrated reduction in drug pressure could stabilize the evolution and the pathogenic potential of resistant virus.

A prospective pilot study was conducted in patients receiving protease inhibitor-based HAART with a resistance genotype predicting less than two active drugs according to the 2002 ANRS algorithm, CD4 counts over or equal to 100/mm3 and plasma HIV RNA below or equal to 5 log/ml. The treatment was low-dose IDV/RTV (200/100 BID) and 3TC 150mg BID. IDV doses were adjusted at week 4 to ensure a Cmin of 250+/-100ng/ml, which, based on a panel of multi-PI resistant viruses, was calculated to yield an inhibitory quotient (Cmin/IC50) of 0.50. Primary end-points were over 25% decrease in CD4 counts (immunological failure-IF), or over 0.7 log increase in plasma HIV RNA (virological failure-VF) at two consecutive monthly visits during the 24-week study. Inclusions were to stop when the total number of failures (VF+IF) reached 7

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection confirmed by Western Blot
* Karnofsky score over or equal to 70
* CD4 over or equal to 200/mm3
* Plasma viral RNA over or equal to 10 000 copies/ml and below 100 000 copies/ml.
* Stability of plasma viral load and CD4-during the last 3 months
* failure of two antiretroviral regimens with 2 PI and one NNRTI
* New efficacy drug on genotype not available
* Treatment on hand with 3 antiretroviral drugs with one PI since 3 months.
* Written inform consent
* Pregnancy

Exclusion Criteria:

* Hemoglobin below 8g/dL
* Neutrophils below 750/mm3
* ASAT, ALAT over 5N
* Hepatic insufficiency (prothrombin below 50%)
* Acute opportunistic infection
* Immunotherapy
* Treatment with active antiretroviral regimen
* Treatment with enzyme inductor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-02; Study Completion 2003-08

PRIMARY OUTCOMES:
Decrease over 25% in CD4 counts (immunological failure-IF), or increase over 0.7 log in plasma HIV RNA (virological failure-VF) at two consecutive monthly visits during the 24-week study

SECONDARY OUTCOMES:
Development of an HIV-1-related AIDS defining event
Death
Change in CD4 cell count between baseline and week 24
Change in plasma HIV-RNA level between baseline and week 4, week 8, week 12 and week 24
Change in genotypic and phenotypic resistance between baseline and week 2

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, Principal Investigator — Hopital Avicenne,Bobigny, Service de Médecine Interne; Dominique Costagliola, Study Chair — Inserm U720
Locations (1):
- Service de Medecine Interne hopital Avicenne, Bobigny, France